CLINICAL TRIAL: NCT05079958
Title: Effects of Cognitive-behavioral Education and Exercise Interventions on Smoking Cessation and Physical and Mental Health in Patients With Coronary Heart Disease: Application of the Transtheoretical Model
Brief Title: Effects of Cognitive-behavioral Education and Exercise Interventions on Smoking Cessation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cathay General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CGH-OP108004
Record Dates: First submitted 2021-08-02; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease; Smoking Cessation
Keywords: Coronary artery disease; Trans-theoretical Model; Smoking cessation
MeSH Terms: conditions — Coronary Artery Disease; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: For the third stage, subjects will be recruited and randomly divided into experimental or control group to identify the effect of a 12-week brisk walking on improving the participants' immediate (short-term), three-month, and six month (long-term) health status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage2 - cognitive-behavioral education (Experimental): A quasi-experimental design will be used to determine the effects of a four-week cognitive-behavioral education course related to smoking cessation on the participants' smoking cessation behavior, smoking decision-making, and self-efficacy in smoking cessation.
  Interventions: Behavioral: cognitive-behavioral education
- Stage 3- 12-week brisk walking (Experimental): Subjects who are at the "preparation " and "action" stage will be recruited and randomly divided into experimental or control group to identify the effect of a 12-week brisk walking on improving the participants' immediate (short-term), three-month, and six month (long-term) health status.
  Interventions: Behavioral: 12-week brisk walking

INTERVENTIONS:
Behavioral: cognitive-behavioral education — four-week cognitive-behavioral education course
  Arms: Stage2 - cognitive-behavioral education
Behavioral: 12-week brisk walking — 12-week brisk walking
  Arms: Stage 3- 12-week brisk walking

SUMMARY:
The purpose of the study is to adopt the Trans-theoretical Model to facilitate step-by-step changes in a patient's smoking behavior and explore the effect of "Cognitive-Behavioral Education Course" and "Exercise Program" on Smoking cessation, physical health, and mental health of smokers with CAD.

DETAILED DESCRIPTION:
Smoking is a major risk factor of coronary artery disease (CAD) and is responsible for the death of one in three patients with cardiovascular diseases. Smoking cessation is one of the most favorable methods for reducing the risk of cardiovascular diseases; even for patients with a heart disease, quitting smoking can reduce the chance of a relapse of said disease. However, the Health Promotion Administration revealed that among male patients with acute myocardial infarction (AMI), 79.5% had smoked and 35.6% continued to smoke after an episode of AMI. Although previous studies confirmed that health education and exercises can increase smoking cessation rates, patients' lack of motivation to quit smoking has resulted in a failure rate of 65.5%. Therefore, identifying methods to strengthen patients' motivation to quit smoking is a key to successfully achieving smoking cessation.

The purpose of the study is to adopt the Trans-theoretical Model to facilitate step-by-step changes in a patient's smoking behavior and explore the effect of "Cognitive-Behavioral Education Course" and "Exercise Program" on Smoking cessation, physical health, and mental health of smokers with CAD. This study is composed of three stages in three years period, recruiting patients (who meet the selection criteria) from the cardiology department of a medical center in northern Taiwan. For the first stage, a cross-sectional method will be employed to investigate the relationship between smoking status and various physiological and psychological indicators in patients with CAD. For the second stage, subjects who are at the smoking cessation stage of "precontemplation" and "contemplation" will be recruited.

A quasi-experimental design will be used to determine the effects of a four-week cognitive-behavioral education course related to smoking cessation on the participants' smoking cessation behavior, smoking decision-making, and self-efficacy in smoking cessation. For the third stage, subjects from Stages 1 and 2 who are at the "preparation " and "action" stage will be recruited and randomly divided into experimental or control group to identify the effect of a 12-week brisk walking on improving the participants' immediate (short-term), three-month, and six month (long-term) health status. The primary indicator used for health status evaluation is smoking cessation success rate; the secondary indicators used are physiological status (i.e., nicotine addiction, lung carbon monoxide concentration, heart rate variability, and smoking withdrawal syndrome) and psychological status (i.e., depression and resilience). SPSS for Window 24.0 software will be used in statistical analysis. The type one error is 0.05. In inferences analysis, chi-square test, Pearson correlation coefficient, independent t test, one-way ANOVA and post hoc comparison (scheffe) test will be used to examine the variance among groups. Finally, ANCOVA and GEE mode will be used to test the effectiveness of intervention at stage 1 and stage 2, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Those who meet the diagnosis and can perform aerobic exercise after being referred by a physician.
2. Those who have a clear consciousness and have no mental disorders as recorded in medical records or verbally.
3. Those who can walk on their own.
4. Participated in the first or second phase of the study and the smoking cessation phase is in the preparation and action phases

Exclusion Criteria:

1. Irregular heart rhythm.
2. Install a heart regulator.
3. Those who already have regular exercise (3 times a week, 20-30 minutes of physical activity each time).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Stage3-The change of smoking cessation success rate | 12-weeks, three-month, and six month
  smoking cessation success
Stage2-The change of smoking cessation behavior | Before, 4-weeks.
  Only one question, "Are you currently considering quitting smoking?" The smoking cessation behavior change stage is divided into 5 periods according to the cross-theoretical model, and they are respectively 1. Unintentional period: current smoking, and no smoking cessation will be considered in the next six months. 2. Intent period: currently smoking, but considering quitting in the next six months. 3. Preparation period: currently smoking, and plan to quit smoking within the nearest month. 4. Action period: I have quit smoking, but less than six months. 5. Maintenance period: I have quit smoking for more than six months.

SECONDARY OUTCOMES:
Stage3-The change of Fagerstrom Test for Nicotine Dependence (FTND) | 12-weeks, three-month, and six month
  Used the "Fagerstrom Test for Nicotine Dependence" (FTND) translated by Health Promotion Administration, Ministry of Health and Welfare. The content of the scale includes six questions. The total score of the scale is 0-10 points. The higher the score, the higher the nicotine dependence index; the lower than 4 points means the degree of addiction is not high. If you are determined to quit smoking, you will be successful; 4-6 is divided into addiction High degree, need to work hard to quit smoking; 7-10 points nicotine addiction is very high, and professionals are needed to help quit smoking
Stage3-The change of lung carbon monoxide concentration | 12-weeks, three-month, and six month
  physiological status
Stage3-The change of heart rate variability | 12-weeks, three-month, and six month
  physiological status
Stage3-The change of smoking withdrawal syndrome | 12-weeks, three-month, and six month
  We used French Minnesota Nicotine Withdrawal Scale, MNWS to assess smoking addiction and withdrawal symptoms. This Includes 1 craving for smoking and 8 withdrawal symptoms (depressed mood; irritability, frustration or anger; anxiety; difficulty concentrating; restlessness; increased appetite; difficulty falling asleep; restless sleep and the urge to smoke). The items are the feelings of those who quit smoking in the past day, and are scored on a scale of 0 to 4. Not at all: 0 points; mild: 1 point; moderate: 2 points; quite severe: 3 points; extremely severe: 4 points. The score includes the smoking craving degree and the eight withdrawal symptoms, which are used to evaluate smoking cessation After the impact, the higher the score, the more severe the withdrawal symptoms.
Stage3-The change of the Center for Epidemiological Studies -Depression Scales (CESD-10) | 12-weeks, three-month, and six month
  We used the Center for Epidemiological Studies -Depression Scales (CESD-10). There are a total of 10 questions, measuring the frequency of depression symptoms in the subject within a week. Each item is given a score of 0 to 3, with a total score of 0 to 30. The higher the score, the more severe the depression. When the scale score ≥ 10 points, it indicates that there is a tendency to depression.
Stage3-The change of Taiwanese Version of the Brief Resilience Scale | 12-weeks, three-month, and six month
  We used Taiwanese Version of the Brief Resilience Scale (BRS). The scale has 6 items divided into two dimensions: resilience and succumbing. Questions 1, 3, and 5 are positive questions, the measurement aspect is resilience, questions 2, 4, and 6 are negative questions, and the measurement aspect is yield. The scoring method uses Likert's 5-point scoring method, from 1 to 5 points each representing "strongly disagree" to "strongly agree", and the negative questions are scored in reverse. The BRS score calculation method is to calculate the average of the individual scores of the 6 items. The higher the average, the higher the psychological resilience, and vice versa, the lower the psychological resilience.
Stage2- smoking decision-making | Before, 4-weeks.
  This scale was developed by Chia et al (2013). There are 6 questions on the scale, including "benefits" and "costs". The score for the benefit part is 3-15 points, the higher score indicates that smoking is important, which means that smoking can gain benefits, and smoking is actually bad [negative reaction]. The score for the costs part is scored 3-15 points. The higher the score indicates that smoking will pay the price, meaning that it is important not to smoke [positive reaction].
Stage2- self-efficacy in smoking cessation | Before, 4-weeks.
  The self-efficacy in smoking cessation developed by Ou, Li and Yan (2000).It was used to evaluate the confidence of the subjects to not smoke in various situations. There are a total of 14 questions on the scale. The Likert four-point calculation is used. The scoring method is used to answer that I will never smoke (4 points), I may not smoke (3 points), I may smoke (2 points), and I will definitely smoke (1 point). The score ranges from 14 to 56 points. The higher the score, the better the self-efficacy of refusal to smoke.

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Chun Wei, Principal Investigator — Cathay General Hospital
Locations (1):
- Cathay General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abrantes AM, Farris SG, Minami H, Strong DR, Riebe D, Brown RA. Acute Effects of Aerobic Exercise on Affect and Smoking Craving in the Weeks Before and After a Cessation Attempt. Nicotine Tob Res. 2018 Apr 2;20(5):575-582. doi: 10.1093/ntr/ntx104. PMID 28505303

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT05079958/Prot_SAP_000.pdf